CLINICAL TRIAL: NCT03713996
Title: Insomnia and Type 2 Diabetes: Measurement, Impact and Intervention
Brief Title: The Effect of Cognitive Behavioral Therapy for Insomnia on Type 2 Diabetes Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Patricia Kluding, PhD, Professor and Chair, Department of Physical Therapy and Rehabilitation Science, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00142985
Record Dates: First submitted 2018-10-11; First posted 2018-10-22 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Type2 Diabetes; Insomnia
Keywords: Cognitive Behavioral Therapy for Insomnia; Self-Care; Fatigue; Diabetes; Glycemic Control
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue; Diabetes Mellitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I intervention (Experimental): The intervention includes several face-to-face interview techniques: sleep restriction therapy, stimulus control procedures, sleep hygiene, relaxation training and cognitive components.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- Diabetes Education (Active Comparator): Sleep hygiene, foot care, causes and diagnosis of diabetes, healthy diet, and physical activity will be delivered for the Health Education group. During all sessions, subjects will be encouraged to engage in the discussion through open questions about their experience in diabetes, lifestyle, and understanding about provided materials.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — CBT-I is designed to change sleep habits as well as direct misconceptions about sleep and insomnia. Participants will receive several face-to-face interview techniques: sleep restriction therapy, stimulus control procedures, sleep hygiene, relaxation training and cognitive components. The intervention will be provided in 6-session (one session/week).
  Arms: CBT-I intervention
Other: Health Education — Participants in this arm will receive education in sleep hygiene, foot care, causes and diagnosis of diabetes, healthy diet, and physical activity. The education will be provided in 6-session (1 session/week).
  Arms: Diabetes Education

SUMMARY:
Insomnia is a common sleep disorder, with three main symptoms: difficulty in initiating sleep, difficulty in maintaining sleep, and/or waking up early without ability to return to sleep. Insomnia can contribute to metabolic dysfunction, which can lead to type 2 diabetes (T2D). Diabetes self-care behavior (DSCB) is important in attaining and maintaining glycemic control, which worsens as a result of fatigue. People with insomnia usually suffer from fatigue and inconstant sleep schedule, which negatively influence quality of life. However, the additive effect of behavioral sleep intervention on diabetes outcomes and health status in people with T2D is unknown. Therefore, The overall purpose of this study is to investigate the impact of both insomnia symptoms and CBT-I on people with T2D. The central hypotheses are that people with T2D and insomnia symptoms will have worse sleep, diabetes measures and self-reported outcomes compared to people with T2D only, which might be adjusted with CBT-I.

DETAILED DESCRIPTION:
Insomnia is a common sleep disorder, with three main symptoms: difficulty in initiating sleep, difficulty in maintaining sleep, and/or waking up early without ability to return to sleep. Insomnia can contribute to metabolic dysfunction, which can lead to type 2 diabetes (T2D). Diabetes self-care behavior (DSCB) is important in attaining and maintaining glycemic control, which worsens as a result of fatigue. People with insomnia usually suffer from fatigue, which negatively influences quality of life. However, the additive effect of insomnia symptoms on diabetes outcomes and health status in people with T2D is unknown. Therefore, it is imperative to investigate the contributing factor that affects DSCB and health outcomes to help individuals with diabetes reach their goals.

Assessing sleep variability is very important clinically and practically for people with insomnia. People with insomnia have higher night to night sleep variability compared to healthy individuals. Compared to other populations, people with T2D might suffer from sleep disturbances due to diabetes symptoms such as frequency nocturnal urination, hyperglycemia, insulin resistance, obesity, pain and fatigue, which might influence the sleep variability. The nature of insomnia is not representable by using mean values, as the reduction in the sleep variability values is a predictor for insomnia and depression recovery. Therefore, understanding the sleep variability in people with T2D with or without insomnia symptoms may add complementary evidence for future studies.

An effective treatment for people with insomnia is Cognitive Behavioral Therapy for Insomnia (CBT-I). CBT-I is superior to sleep medications in terms of cost and long term benefits. Although there is currently limited evidence about the effect of CBT-I on people with T2D, CBT-I is a potentially effective intervention given insomnia's relationship with glucose metabolism. The overall purpose of this study is to investigate the impact of both insomnia symptoms and CBT-I on people with T2D. The central hypotheses are that people with T2D and insomnia symptoms will have worse sleep, diabetes measures and self-reported outcomes compared to people with T2D only, which might be adjusted with CBT-I.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 to 75 years
* Self-reported diagnosis of type 2 diabetes
* Insomnia Severity Index >10 and self-reported symptoms of insomnia at least 3 nights/week for the past 3 months for insomnia and type 2 diabetes group
* Insomnia Severity Index ≤10 for type 2 diabetes only group
* Able to attend 6 sessions
* Able to understand and follow verbal commands in English
* Able to travel to our lab

Exclusion Criteria:

* Self-reported neurological diseases (e.g. Alzheimer's disease, Parkinson's disease, Traumatic Brain Injury, Stroke, Multiple Sclerosis)
* Stop-Bang > 4 indicating severe risk of sleep apnea
* Failure to pass Restless Leg Syndrome Diagnostic Index
* Severe pain ≥ 7 out of 10 on Brief Pain Inventory
* Severe symptom level of depression scores ≥ 21 on Beck Depression Inventory
* Severe symptom level of anxiety scores ≥ 15 on Generalized Anxiety Scale-7
* Pregnant women
* Self-reported following medical issues: Chronic Fatigue Syndrome, Fibromyalgia, and Rheumatic Diseases
* Speech deficits or significant auditory impairment
* Night-shift work
* Self-reported Bipolar and Seizure Disorders
* Heavy alcohol drinker (≥15 drinks per week for men and ≥ 8 drinks per week for women)
* Dialysis/blindness/trans-femoral amputation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Insomnia severity will be assessed at the baseline and 8 weeks.
  The Insomnia Severity Index is a self-report measure designed to evaluate the nature, severity, and impact of insomnia.Seven-items assess severity of sleep onset, sleep maintenance, early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress due to the sleep difficulties.This is self-reported seven items on a five-point Likert scale from zero (not at all satisfied) to four (very much satisfied). Total scores range from 0 to 28, with higher scores indicating greater insomnia severity.

SECONDARY OUTCOMES:
Change in the Variability of Total Sleep Time in Minutes using Objective Measure, Actigraph | The variability of total sleep time for 7 nights will be assessed at the baseline and 8 weeks.
  Actigraph is a useful measure for common sleep parameters including total in minutes being awake, total sleep time, sleep latency, and sleep efficiency. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of total sleep time (in minutes) divided by the mean of 7 nights of total sleep time (in minutes) multiply by 100). The range of Total Sleep Time variability is from 0% to 100%, with higher score indicating higher variability of Total Sleep Time.
Change in the Variability of Wake after Sleep Onset in Minutes using Objective Measure, Actigraph | The variability of wake after sleep onset for 7 nights will be assessed at the baseline and 8 weeks.
  Actigraph is a useful measure for common sleep parameters including total in minutes being awake, total sleep time, sleep latency, and sleep efficiency. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of total Wake after Sleep Onset (in minutes) divided by the mean of 7 nights of total Wake after Sleep Onset (in minutes) multiply by 100). The range of Wake after Sleep Onset variability is from 0% to 100%, with higher score indicating higher variability of Wake after Sleep Onset.
Change in the Variability of Sleep Latency in Minutes using Objective Measure, Actigraph | The variability of sleep latency for 7 nights will be assessed at the baseline and 8 weeks.
  Actigraph is a useful measure for common sleep parameters including total in minutes being awake, total sleep time, sleep latency, and sleep efficiency. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of total sleep latency (in minutes) divided by the mean of 7 nights of total sleep latency (in minutes) multiply by 100). The range of Sleep Latency variability is from 0% to 100%, with higher score indicating higher variability of Sleep Latency.
Change in the Variability of Sleep Efficiency using Objective Measure, Actigraph | The variability of sleep efficiency for 7 nights will be assessed at the baseline and 8 weeks.
  Actigraph is a useful measure for common sleep parameters including total in minutes being awake, total sleep time, sleep latency, and sleep efficiency. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of sleep efficiency (in percentage) divided by the mean of 7 nights of sleep efficiency (in percentage) multiply by 100). The range of Sleep Efficiency variability is from 0% to 100%, with higher score indicating higher variability of Sleep Efficiency.
Change in the Variability of Total Sleep Time in Minutes using Subjective Measure, Sleep Diary | The variability of total sleep time for 7 nights will be assessed at the baseline and 8 weeks.
  Sleep diary is a subjective gold stander sleep measures. Subjects will be asked to report their daily sleep including time in bed and out of bed, total sleep time, number of awakening and total time being awake. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of total sleep time (in minutes) divided by the mean of 7 nights of total sleep time (in minutes) multiply by 100). The range of Total Sleep Time variability is from 0% to 100%, with higher score indicating higher variability of Total Sleep Time.
Change in the Variability of Wake after Sleep Onset in Minutes using Subjective Measure, Sleep Diary | The variability of wake after sleep onset for 7 nights will be assessed at the baseline and 8 weeks.
  Sleep diary is a subjective gold stander sleep measures. Subjects will be asked to report their daily sleep including time in bed and out of bed, total sleep time, number of awakening and total time being awake. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of total Wake after Sleep Onset (in minutes) divided by the mean of 7 nights of total Wake after Sleep Onset (in minutes) multiply by 100). The range of Wake after Sleep Onset variability is from 0% to 100%, with higher score indicating higher variability of Wake after Sleep Onset.
Change in the Variability of Sleep Latency in Minutes using Subjective Measure, Sleep Diary | The variability of sleep latency for 7 nights will be assessed at the baseline and 8 weeks.
  Sleep diary is a subjective gold stander sleep measures. Subjects will be asked to report their daily sleep including time in bed and out of bed, total sleep time, number of awakening and total time being awake. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of total sleep latency (in minutes) divided by the mean of 7 nights of total sleep latency (in minutes) multiply by 100). The range of Sleep Latency variability is from 0% to 100%, with higher score indicating higher variability of Sleep Latency.
Change in the Variability of Sleep Efficiency using Subjective Measure, Sleep Diary | The variability of sleep efficiency for 7 nights will be assessed at the baseline and 8 weeks.
  Sleep diary is a subjective gold stander sleep measures. Subjects will be asked to report their daily sleep including time in bed and out of bed, total sleep time, number of awakening and total time being awake. Sleep efficiency will be calculated based on the ratio of total sleep time and total time in bed multiply by 100. The variability of 7 nights will be measured by Coefficient of Variance (standard deviation of 7-nights of sleep efficiency (in percentage) divided by the mean of 7 nights of sleep efficiency (in percentage) multiply by 100). The range of Sleep Efficiency variability is from 0% to 100%, with higher score indicating higher variability of Sleep Efficiency.
Change in Fatigue Severity Scale Total Score | Fatigue severity will be assessed at the baseline and 8 weeks.
  Fatigue Severity Scale is a validated 9-item questionnaire, to assess the fatigue in daily life and differentiate between fatigue and clinical depression. Total scores in which < 4 indicate no fatigue, scores between 4 and 4.9 indicate moderate fatigue, and score >5 indicate severe fatigue. The mean score of the nine items will be used, which ranges from 1 to 7.
Change in Diabetes Self-Care Behavior using Diabetes Care Profile | Change in each sub-scale on the Diabetes Care Profile from the baseline and at 8 weeks
  Diabetes care profile is a validated instrument that measures self-reported diabetes control, psychological and social factors including Control Problems, Social and Personal Factors, Negative Attitude, Positive Attitude, Self-Care Adherence, and Diet Adherence. Each item on the Diabetes Care Profile is rated on 1 to 5 scales to evaluate the frequency of symptoms. Control Problems, Social and Personal Factors, and Negative Attitude are rated on a scale where 1 is good and 5 is poor; Positive Attitude, Self-Care Adherence, and Diet Adherence are rated on a scale where 5 is good and 1 is poor. Each sub-scale will represent an aspect in the diabetes self-care behavior.
Change in Glycemic Control Level | A1C will be assessed at the baseline and 8 weeks.
  Glycemic control will be tested using HbA1c testing Kit. HbA1c indicates the average blood glucose level of people with diabetes over the previous 2-3 months. Higher score on the A1C indicates poor glycemic control
Change in Epworth Daytime Sleepiness Scale Total Score | Daytime sleepiness will be assessed at the baseline and 8 weeks.
  The Epworth Sleepiness Scale will be utilized to evaluate the daytime sleepiness and subjectively investigate the likelihood of unintentionally falling asleep or increased difficulty in staying awake . It encompasses 8 items where the subjects rate how likely they would be to fall asleep in 8 different states of daily activities. A 4-point Likert scale ranging between 0 "never doze" and 3 "high chance of dozing". Total score will be used, which ranges from 0 to 24.
Change in The Pittsburgh Sleep Quality Index Global Score | Sleep quality will be assessed at the baseline and 8 weeks.
  The Pittsburgh Sleep Quality Index is a validated 19-item questionnaire, and it differentiates between poor sleepers and good sleepers. it is derived from 7 items including perceived sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. These items are separately scored from 0-3, with 3 representing the negative extreme, and summed to provide a global score. The total score of Pittsburgh Sleep Quality Index will be used, which ranges from 0 to 21. Higher scores indicate poor sleep quality.
Change in Random Glucose Level | Random glucose level will be assessed at the baseline and 8 weeks.
  Glucose meter will be utilized to assess the glucose level.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The protocol of this study will be published. We already submit the protocol to an Open access journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The protocol will be submitted to an open access journal and will be available to everyone.

REFERENCES:
- [Derived] Alshehri MM, Alothman SA, Alenazi AM, Rucker JL, Phadnis MA, Miles JM, Siengsukon CF, Kluding PM. The effects of cognitive behavioral therapy for insomnia in people with type 2 diabetes mellitus, pilot RCT part II: diabetes health outcomes. BMC Endocr Disord. 2020 Sep 5;20(1):136. doi: 10.1186/s12902-020-00612-6. PMID 32891140
- [Derived] Alshehri MM, Alenazi AM, Hoover JC, Alothman SA, Phadnis MA, Rucker JL, Befort CA, Miles JM, Kluding PM, Siengsukon CF. Effect of Cognitive Behavioral Therapy for Insomnia on Insomnia Symptoms for Individuals With Type 2 Diabetes: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2019 Dec 19;8(12):e14647. doi: 10.2196/14647. PMID 31855189